CLINICAL TRIAL: NCT04458012
Title: Epidemiological Study of Dry Eye Disease in Stavanger: Dry Eye Disease in Patients With Age-related Macular Degeneration Treated With Intravitreal Injections
Brief Title: Epidemiological Study of Dry Eye Disease in Stavanger: Dry Eye Disease in Patients Treated With Intravitreal Injections
Acronym: EPISTA1
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Tor Paaske Utheim (Unknown); Vegard Asgeir Forsaa (Unknown); Vilde Marie Thomseth (Unknown)
Responsible Party: Principal Investigator, Agni Malmin, MD, Helse Stavanger HF
Other Study IDs: EPISTA1
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-06

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tear fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Oculus Keratograph. Schirmer test. Tear fluid sample. — Objective measurements of the ocular surface using Oculus 5 keratograph. Slit lamp examination and tear fluid sample using Schirmer strips.

SUMMARY:
To investigate prevalence of dry eye disease in Norwegian patients with age-related macular degeneration receiving intravitreal injections, as well as to reveal possible risk factors of DED in this population.

DETAILED DESCRIPTION:
Questionaires (OSDI, McMonnies) and clinical investigation using the Oculus 5 Keratograph for objective ocular surface evaluation. Tear fluid samples will be collected for later biochemical analysis.

ELIGIBILITY:
Inclusion Criteria:

* AMD diagnosis
* Treated with intravitreal injection agents

Exclusion Criteria:

* Not able to cooperate

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age related macular degeneration receiving intravitreal injections with anti-vegf.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-25 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Dry eye disease in patients receiving intravitreal injections | 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Stavanger University Hospital, Department of Ophthalmology, Stavanger, Norway

IPD SHARING:
Plan to Share IPD: No